CLINICAL TRIAL: NCT06243731
Title: Retrospective Chart Review of Safety Outcomes Associated With Use of Maribavir in Patients With Post-transplant Refractory Cytomegalovirus (CMV) Infection and Comorbid Severe Chronic Kidney Disease (CKD) or Comorbid End-stage Renal Disease (ESRD), Including Patients on Peritoneal Dialysis or Hemodialysis
Brief Title: A Study of Maribavir in Adults With Kidney Failure Who Have a Cytomegalovirus (CMV) Infection After Transplantation
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-4007; EUPAS1000000006 (Registry Identifier: EUPAS)
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cytomegalovirus (CMV); Kidney Disease; Kidney Failure
Keywords: Drug therapy
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants With Kidney Failure: The study cohort will comprise of participants aged 18 years or older treated with maribavir for a refractory CMV infection and who have severe CKD or comorbid ESRD including participants on peritoneal dialysis or hemodialysis. Data from eligible participants will be assessed from index date (Day 0: the day of initiation of the first maribavir treatment course during the eligibility period) until 7 days after the date of the end of supply of the last prescription of treatment or date of death or end of data availability, or treatment completion/discontinuation whichever occurs first.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to assess the safety of maribavir in adults with severe CKD or comorbid ESRD including participants on artificial filtering of the kidney (dialysis) or the blood (hemodialysis).

In this study, already existing data will be collected from the participant's medical records. The study will only review data collected as part of the normal clinical routine and will not impact the standard medical care and treatment of participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults more than and equal to (≥) 18 years of age at index date.
* Diagnosis of comorbid ESRD or comorbid severe CKD prior to the index date.

  * If ESRD (including participants on peritoneal dialysis or hemodialysis): participant diagnosed with ESRD confirmed by an estimated glomerular filtration rate (eGFR) less than (<) 15 milliliters per minute per 1.73 square meters (mL/min/1.73m^2).
  * If severe CKD: participant diagnosed with severe CKD confirmed by an eGFR of 15 to <30 mL/min/1.73m^2 at index.
* Participant has undergone solid organ transplant (SOT) or hematopoietic stem cell transplantation (HSCT) before index date.
* Participant was diagnosed with refractory (with or without resistance) CMV during the latest post-transplant period.
* Participant initiated treatment with maribavir in routine practice within the eligibility period and received at least 1 dose of maribavir.
* Informed consent provided (where required by local regulations) before data collection commences.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants treated with maribavir for a refractory (with or without resistance) CMV infection and who have severe CKD or comorbid ESRD including participants on peritoneal dialysis or hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Time from index treatment date until 7 days after the date of the end of supply of the last prescription of treatment or date of death, whichever occurs first (up to 4 years)
  An AE is defined as any untoward medical occurrence (including a symptom or disease or an abnormal laboratory finding) in a participant or clinical investigation participants administered a medicinal product and which does not necessarily have a causal relationship with the treatment. A serious adverse event (SAE) is any event that results in: death; life-threatening event; requires inpatient hospitalization or results in prolongation of existing hospitalization; persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or a medically important event.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events of Special Interest (AESIs) | Time from index treatment date until 7 days after the date of the end of supply of the last prescription of treatment or date of death, whichever occurs first (up to 4 years)
  An AESI is defined as AEs that will be specifically highlighted to the Investigator. AESIs are as follows: Immunosuppressant drug concentration level increased, tissue-invasive CMV disease, relapse or progression of the underlying disease for which the transplant was performed, taste disturbance (dysgeusia), Nausea, vomiting, diarrhea, invasive fungal or bacterial infections, graft-versus-host-disease (GVHD), leukopenia including neutropenia, lymphocytopenia, and low white blood cell (WBC) count, anemia including low hemoglobin and thrombocytopenia including low platelets count.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (25):
- Belgium (2):
  - Hopital Erasme - PPDS, Anderlecht, Brussels Capital
  - UZ Leuven - PPDS, Leuven, Vlaams Brabant
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn, Harju
  - Tartu University Hospital, Tartu
- France (5):
  - CHU de Brest - Hopital La Cavale Blanche, Brest, Finistere
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux, Gironde
  - CHU de Montpellier - Hopital Lapeyronie, Montpellier, Herault
  - CHU de Grenoble Alpes - Hopital Michallon, La Tronche, Isere
  - AP-HP - Hopital Henri Mondor, Créteil, Val-de-Marne
- Germany (2):
  - Universitatsklinikum Wurzburg, Würzburg, Bavaria
  - Universitatsklinikum Leipzig, Leipzig, Saxony
- Italy (2):
  - Azienda Ospedaliera Dei Colli - Ospedale Monaldi, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Spain (8):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga Hospital General, Málaga
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- United Kingdom (4):
  - Dorset County Hospital, Dorchester, Dorset
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - King's College Hospital, London
  - Wrexham Maelor Hospital, Wrexham

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/562b008bd1aa4302?idFilter=%5B%22TAK-620-4007%22%5D